CLINICAL TRIAL: NCT07258290
Title: Safety and Clinical Performance of the Drug Eluting Resorbable Coronary Magnesium Scaffold System (Freesolve) in the Treatment of Subjects With de Novo Lesions in Native Coronary Arteries
Brief Title: Safety and Clinical Performance of the Freesolve Resorbable Magnesium Scaffold (RMS) System in Subjects With Coronary Artery Lesions
Acronym: BIOMAG-III
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Teleflex (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: G230176
Record Dates: First submitted 2025-11-20; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Coronary Disease; Heart Diseases; Cardiovascular Diseases; Arteriosclerosis; Arterial Occlusive Diseases; Vascular Diseases; Chest Pain; Pain; Neurologic Manifestations; Signs and Symptoms; Pathological Conditions, Signs and Symptoms; Coronary Artery Disease; Myocardial Ischemia; Acute Coronary Syndrome; Angina Pectoris
Keywords: Resorbable Magnesium Scaffold; Sirolimus; RMS; Drug eluting absorbable metal scaffold
MeSH Terms: conditions — Coronary Disease; Heart Diseases; Cardiovascular Diseases; Arteriosclerosis; Arterial Occlusive Diseases; Vascular Diseases; Chest Pain; Pain; Neurologic Manifestations; Signs and Symptoms; Pathological Conditions, Signs and Symptoms; Coronary Artery Disease; Myocardial Ischemia; Acute Coronary Syndrome; Angina Pectoris

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Freesolve RMS (Experimental): Intervention with a Freesolve Sirolimus Eluting Coronary Resorbable Magnesium Scaffold (RMS) System
  Interventions: Device: Freesolve RMS
- Xience DES (Active Comparator): Intervention with a Xience Everolimus Eluting Stent System
  Interventions: Device: Xience DES

INTERVENTIONS:
Device: Freesolve RMS — Freesolve Sirolimus-Eluting Coronary Resorbable Magnesium Scaffold (RMS) System, a drug-eluting balloon-expandable resorbable scaffold
  Arms: Freesolve RMS
Device: Xience DES — Xience Everolimus Eluting Stent System
  Arms: Xience DES

SUMMARY:
The objective of this study is to assess the safety and efficacy of the Freesolve resorbable magnesium scaffold (RMS) in the treatment of subjects with up to two de novo lesions in native coronary arteries compared to the Xience coronary drug-eluting stent (DES) system

DETAILED DESCRIPTION:
The BIOMAG-III clinical trial is a prospective, international, multi-center, single-blinded, randomized controlled, non-inferiority trial to compare the Freesolve Sirolimus Eluting Coronary Resorbable Magnesium Scaffold (Freesolve RMS) System with the Xience Everolimus Eluting Stent (Xience DES) System. with respect to Target Lesion Failure (TLF) rate at 12 months. Subjects will be randomized in a 2:1 fashion Freesolve to Xience. A total of up to 1859 subjects will be randomized at up to 120 total sites worldwide including North America, Europe, and Asia Pacific. Clinical follow-up will be conducted at 1, 6, and 12 months and at 2, 3, 4, and 5 years post-procedure.

ELIGIBILITY:
Clinical Inclusion Criteria:

1. Subject is ≥ 18 years and ≤ 80 years of age
2. Subject has provided written informed consent as approved by the Ethics Committee / Institutional Review Board (IRB) of the respective clinical site prior to the study related procedures
3. Subject is eligible for PCI according to the applicable guidelines
4. Subject is an acceptable candidate for coronary artery bypass surgery
5. Subjects with stable or unstable angina pectoris, documented silent ischemia/abnormal physiologic testing or hemodynamically stable non-ST elevation myocardial infarction (NSTEMI) patients without angiographic evidence of thrombus at target lesion

   Note: STEMI patients may be eligible for the study for treatment of selected non-culprit lesions, if:
   * Subject and target lesion(s) meet all inclusion and no exclusion criteria and consent occurs at least ≥ 72 hours after successful treatment of the culprit lesion(s) [lesion(s) causing the acute STEMI];
   * Subject is hemodynamically stable with documented declining cardiac biomarkers;
   * Target lesion(s) to be treated are not located in the culprit vessel(s) and are not culprit lesion(s)
6. Subject is eligible for Dual Antiplatelet Therapy (DAPT) with aspirin plus either clopidogrel, prasugrel, ticagrelor or ticlopidine
7. Documented left ventricular ejection fraction (LVEF) ≥ 30% within 6 months prior to or during the procedure (prior to randomization)
8. Subject is willing and able to comply with protocol requirements, including completion of study visits for the duration of the study

Angiographic Inclusion Criteria:

1. Subjects with a maximum of two single de novo target lesions each in separate native coronary arteries
2. Target vessel must have a reference diameter between 2.5-4.2 mm by operator visual estimation, which may be assisted by Quantitative Coronary Angiography (QCA) / Intravascular Ultrasound (IVUS) / Optical Coherence Tomography (OCT)
3. Target lesion(s) must be ≤ 36 mm in length by operator visual estimation, which may be assisted by QCA / IVUS / OCT, (or < 20 mm for target lesion(s) to be treated with a study device < 3.0 mm in diameter) and must be amenable to treatment with a single study device
4. Target lesion stenosis ≥ 50% and < 100% by operator visual estimation, which may be assisted by QCA / IVUS / OCT. Target lesion stenosis < 70% by visual estimation, should have clinical justification for treatment as per local standards.
5. Target lesion must have a Thrombolysis in Myocardial Infarction (TIMI) flow ≥ 1

Clinical Exclusion Criteria:

1. Subject is pregnant and/or breastfeeding or intends to become pregnant during the duration of the study
2. Subject has clinical symptoms and/or electrocardiogram (ECG) changes consistent with STEMI < 72 hours prior to the index procedure Note: Hemodynamically stable non-STEMI (NSTEMI) subjects are eligible for study enrollment
3. Subject has undergone prior PCI within the target vessel during the last 12 months prior to the index procedure or prior PCI within a non-target vessel < 72 hours prior to the index procedure
4. Subject is on dialysis or has impaired renal function (serum creatinine > 2.5 mg/dL or 221 µmol/L, determined within 7 days prior to the index procedure)
5. Subject has a known allergy to contrast medium that cannot be adequately premedicated, or any known allergy to aspirin, P2Y12 inhibitors, both heparin and bivalirudin, sirolimus, everolimus (or similar limus drugs), poly L-lactide, the scaffold material (magnesium, aluminum, tantalum), or Xience stent material (cobalt, chromium, tungsten, nickel, methacrylic polymer, and fluoropolymer)
6. Subject is receiving oral or intravenous immunosuppressive therapy (inhaled steroids are permitted) or has known life-limiting immunosuppressive or autoimmune disease (e.g., human immunodeficiency virus, systemic lupus erythematosus; diabetes mellitus is permitted)
7. Life expectancy less than 1 year
8. Planned surgery or dental surgical procedure within 6 months after index procedure, unless DAPT can be maintained
9. In the investigator's opinion subject will not be able to comply with the follow-up requirements
10. Subjects under oral anticoagulation therapy (OAC) prior to index procedure unless DAPT + OAC (i.e., triple therapy) can be maintained for a minimum of 1 month
11. Subject has had a stroke or transient ischemic attack (TIA) within 6 months prior to the index procedure
12. Subject with active bleeding disorder, active coagulopathy, or any other reason, who is ineligible for DAPT
13. Subject is currently participating or plans to participate in another study with an investigational device or an investigational drug
14. Subject has known severe aortic or mitral valve stenosis/insufficiency or has previously undergone transcatheter aortic valve replacement (TAVR)

Angiographic Exclusion Criteria:

1. Target vessel has been previously treated and the target lesion is within 5 mm proximal or distal to the previously treated lesion
2. Left main coronary artery disease
3. Target lesion is totally occluded (100% stenosis)
4. Thrombus in target vessel
5. Future planned staged PCI either in target or non-target vessel
6. Ostial target lesion within the left anterior descending (LAD), left circumflex (LCX), or right coronary artery (RCA) (within 5.0 mm of vessel origin)
7. Target lesion involves a side branch ≥ 2.0 mm in diameter that requires a two-device strategy after pre-dilatation
8. Target lesion is located in or supplied by an arterial or venous bypass graft
9. Target lesion with excessive tortuosity proximal to or within the lesion based on visual estimation or heavily calcified target lesion which cannot be adequately pre-dilated by a non-compliant and/or cutting/scoring balloon as described in angiographic exclusion criteria 10
10. Target lesion requires treatment with a device other than the non-compliant balloon and/or cutting/scoring balloon prior to scaffold/stent placement (including but not limited to atherectomy devices, intravascular lithotripsy, drug-coated balloons, etc.)
11. Target vessel was treated with brachytherapy any time prior to the index procedure.
12. Unsuccessful pre-dilatation, defined as residual stenosis > 20% (by visual estimation) and/or angiographic complications (e.g., distal embolization, side branch closure, flow-limiting dissections)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1859 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2029-06 (Estimated); Study Completion 2033-06 (Estimated)

PRIMARY OUTCOMES:
Target Lesion Failure (TLF) rate at 12 months post-index procedure | 12 months
  The primary endpoint is Target Lesion Failure (TLF) at 12 months, a composite of Cardiac Death, Target Vessel Q-wave or non-Q wave MI, or clinically driven target lesion revascularization (TLR).

SECONDARY OUTCOMES:
Procedure success | Hospital Discharge (6-24 hours post-index procedure)
  Procedure success defined as achievement of < 30% final residual diameter stenosis [by Quantitative Coronary Angiography (QCA) or visual estimation] of the target lesion using the assigned study device only, without the occurrence of cardiac death, Q-wave or non-Q-wave MI, or repeat revascularization of the target lesion during the hospital stay
Device Success | Hospital Discharge (6-24 hours post-index procedure)
  Device Success defined as a final residual diameter stenosis of < 30% by QCA or visual estimation, using the assigned device only with
  * successful delivery of the device to the target lesion, and
  * appropriate device deployment, and
  * successful removal of the delivery system
Target lesion failure (TLF) | Time Frame: 1, 6 months and 2, 3, 4 and 5 years post-index procedure
  TLF is defined as a composite of Cardiac Death, Target Vessel Q-wave or non-Q-wave myocardial infarction (MI), or clinically driven Target Lesion Revascularization (TLR)
Target Vessel Failure (TVF) | 1, 6, 12 months and 2, 3, 4 and 5 years post-index procedure
  Target Vessel Failure (TVF), a composite of Cardiac Death, Target Vessel Q-wave or non-Q wave MI, or clinically driven Target Vessel Revascularization (TVR)
Cardiac death | 1, 6, 12 months and 2, 3, 4 and 5 years post-index procedure
Cardiovascular death | 1, 6, 12 months and 2, 3, 4 and 5 years post-index procedure
All-cause mortality | 1, 6, 12 months and 2, 3, 4 and 5 years post-index procedure
Target vessel MI in accordance with the primary endpoint definitions for periprocedural and non-periprocedural MI | 1, 6, 12 months and 2, 3, 4 and 5 years post-index procedure
Any MI (including non-target vessel territory) | 1, 6, 12 months and 2, 3, 4 and 5 years post-index procedure
Clinically driven TLR | 1, 6, 12 months and 2, 3, 4 and 5 years post-index procedure
Clinically driven TVR | 1, 6, 12 months and 2, 3, 4 and 5 years post-index procedure
Scaffold/stent thrombosis (definite, definite/probable, probable) according to Academic Research Consortium (ARC-2) criteria for acute, sub-acute, late, very late and cumulative scaffold/stent thrombosis | 1, 6, 12 months and 2, 3, 4 and 5 years post-index procedure
Powered Secondary Endpoint 1: TLF from 1-5 Years | 1 to 5 years post-index procedure
  A powered secondary endpoint of cumulative TLF rates between 1 and 5 years post-procedure will be evaluated.
Powered Secondary Endpoint 2: TLF at 12 Months in the Diabetic Population | 12 months post-index procedure
  A powered secondary endpoint of TLF at 12 months in the diabetic population will be evaluated.

IPD SHARING:
Plan to Share IPD: No
No IPD sharing is planned at this time. This study evaluates an investigational device under an FDA IDE. The sponsor may consider sharing de-identified IPD under controlled access following completion of primary endpoint analysis and regulatory review. Summary results will be reported in scientific publications and public registries.